CLINICAL TRIAL: NCT01634685
Title: A Phase I Study of the Phosphatidylserine-Targeting Antibody Bavituximab in Combination With Capecitabine and Radiation Therapy for the Treatment of Stage II and III Rectal Adenocarcinoma
Brief Title: A Phase I Study of Bavituximab, Capecitabine, and Radiation for the Treatment of Rectal Adenocarcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU 032012-025
Record Dates: First submitted 2012-06-28; First posted 2012-07-06 (Estimated); Last update posted 2020-08-20 (Actual); Status verified 2018-05

CONDITIONS: Rectal Adenocarcinoma
Keywords: Rectal cancer; Bavituximab; Capecitabine; Radiation Therapy
MeSH Terms: conditions — Rectal Neoplasms | interventions — Radiation; bavituximab; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bavituximab, Capecitabine, Radiation (Experimental): one arm
  Interventions: Radiation: Radiation; Drug: Bavituximab; Drug: Capecitabine

INTERVENTIONS:
Radiation: Radiation — Radiation therapy will be administered daily, Monday-Friday, for a total of 28 treatments, delivered at 1.8 Gy/fraction.
Drug: Bavituximab — Bavituximab will be delivered concurrently with the radiation therapy for 6 weeks (one time each week), followed by 2 weeks of bavituximab administration by itself.
  Other Names: Phosphatidylserine-Targeting Antibody
Drug: Capecitabine — capecitabine, will be delivered twice daily p.o. on the days of radiation treatment, at a dose of 825 mg/m2.
  Other Names: Xeloda

SUMMARY:
This is a phase I study incorporating bavituximab into the care of patients with rectal adenocarcinoma simultaneously treated with capecitabine and radiation therapy. There is no reference therapy as we are trying to identify the MTD of bavituximab in this combination.

DETAILED DESCRIPTION:
The investigational drug in this protocol is bavituximab, which will be delivered concurrently with the radiation therapy for 6 weeks (one time each week), followed by 2 weeks of bavituximab administration by itself. If the other therapies are terminated after week 4 the bavituximab treatment may be continued per protocol. A chemotherapy agent, capecitabine, will be delivered twice daily p.o. on the days of radiation treatment, at a dose of 825 mg/m2. Radiation therapy will be administered daily, Monday-Friday, for a total of 28 treatments, delivered at 1.8 Gy/fraction. Surgery will follow the last bavituximab administration by 4-8 weeks (6-10 weeks following completion of radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-proven invasive adenocarcinoma of the rectum, stage T3-4 and/or node-positive (AJCC stage II or III). For the purpose of this study, a tumor is located in the "rectum" when its distal edge is located within 12cm of the anal verge. The distal edge of the tumor can be delineated by digital examination or endoscopic examination, including colonoscopy, although rigid proctoscopy is preferred.
* Age > 18 years.
* Performance status of 0 or 1 on the ECOG scale is required (See Appendix 1).
* Adequate organ and marrow function as defined below:

  * leukocytes ≥ 3,000/mcL
  * absolute neutrophil count ≥ 1,500/mcL
  * platelets ≥ 100,000/mcl
  * total bilirubin within normal institutional limits
  * AST(SGOT)/ALT(SGPT) ≤ 2.5 X institutional upper limit of normal
  * creatinine <1.5 X institutional upper limits of normal
  * aPTT ≤1.5 X institutional upper limits of normal
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 90 days following completion of therapy. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* A female of child-bearing potential is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

  * Has not undergone a hysterectomy or bilateral oophorectomy;
  * or has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months).
* Ability to understand and the willingness to sign a written informed consent

Exclusion Criteria:

* Known history of bleeding diathesis or coagulopathy (e.g., von Willebrand disease or hemophilia).
* Bleeding

  1. Clinically significant bleeding, such as gross hematuria, gastrointestinal bleeding (excluding bleeding from rectal tumor), and hemoptysis within the 12 months before screening. If clinically significant bleeding has occurred within 12 months of screening but the cause has been identified and adequately treated (e.g., cystitis, ulcer), then this exclusion criterion does not apply.
  2. Minor biopsy-related bleeding lasting < 24 hours and resolved at least 1 week before Study Day 1 is allowed.
* Venous thromboembolic events (e.g., deep vein thrombosis or pulmonary embolism) within 6 months of screening.
* Ongoing therapy with oral or parenteral anticoagulants; low-dose anticoagulation to maintain patency of lines is allowed.
* Concurrent estrogens, anti-estrogens or progesterone compounds.
* Any prior radiation for rectal cancer.
* Symptomatic or clinically active brain metastases.
* Major surgery within 4 weeks of Study Day 1.
* Pregnant or nursing women.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, history of blood clotting abnormalities, or psychiatric illness/social situations that would limit compliance with study requirements.
* Symptomatic coronary artery disease, cerebrovascular accident, transient ischemic attack, myocardial infarction, or unstable angina pectoris within 6 months of screening.
* Known chronic infection with human immunodeficiency virus (HIV) or viral hepatitis.
* Known hypersensitivity to any components of the treatments.
* History of malignancy other than non-melanoma skin cancers within 5 years prior to study enrollment.
* Subjects receiving other investigational agents thirty days prior to study treatment or during treatment.
* History of inflammatory bowel disease

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2012-08-08 (Actual); Primary Completion 2015-10-30 (Actual); Study Completion 2017-10-06 (Actual)

PRIMARY OUTCOMES:
dose-limiting toxicities (DLT) | 28 days
  To determine dose-limiting toxicities (DLT) for bavituximab when administered on a weekly basis concurrently with external beam radiation therapy.

SECONDARY OUTCOMES:
adverse events | 12 weeks
  To describe the adverse events associated with bavituximab when administered on a weekly basis concurrently with external beam irradiation and capecitabine
MR imaging and histopathological response | 12 weeks
  To describe any preliminary evidence of anti-tumor activity by assessment of objective response as determined by MR imaging and histopathological response in patients with T3-4 and/or node-positive rectal adenocarcinoma.
tumor-vasculature parameters | week 3 and 12
  To determine if the combination of bavituximab, capecitabine, and radiation therapy induces changes in tumor-vasculature parameters as assessed by DCE-MRI, in selected patients.
maximally tolerated dose (MTD) | 28 days
  To determine maximally tolerated dose (MTD) for bavituximab when administered on a weekly basis concurrently with external beam radiation therapy.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No